CLINICAL TRIAL: NCT00916617
Title: A Multicenter, Open Label, Multiple Dose, Parallel Group Investigation Of The Long-term Safety, Tolerability, Reactogenicity, Pharmacokinetics And Pharmacodynamics Of Aab-001 Administered Subcutaneously In Subjects With Mild To Moderate Alzheimer's Disease
Brief Title: Study Evaluating The Long-Term Safety And Efficacy Of Subcutaneous Bapineuzumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated on August 6, 2012, because 2 large Phase 3 studies showed no clinical benefit. This decision was not based on any new safety concerns.
Sponsor: Pfizer (Industry)
Collaborators: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3133L1-2204; B2521009 (Other: Alias Study Number)
Record Dates: First submitted 2009-06-04; First posted 2009-06-09 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-04

CONDITIONS: Alzheimer Disease
Keywords: open-label; safety; antibody
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): 5 mg/week
  Interventions: Drug: bapineuzumab

INTERVENTIONS:
Drug: bapineuzumab — 5 mg/week subcutaneous bapineuzumab

SUMMARY:
This study will evaluate the safety and tolerability of bapineuzumab when administered by subcutaneous injection. The study is open only to subjects who participated in the preceding double-blind study (3133L1-2203 US). Subjects will receive weekly injections of bapineuzumab for 3 years (156 doses). One dosage level will be included: 5 mg/week. All subjects will receive active treatment (bapineuzumab) and no subjects will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer disease
* Completed preceding double-blind study (3133L1-2203 US)
* MMSE score > 9.

Exclusion Criteria:

* Significant brain MRI abnormalities
* Clinically important psychiatric symptoms
* History of stroke

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2009-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Pharmacology Research Institute, Encino, California
  - Brain Matters Research, Delray Beach, Florida
  - MD Clinical, Hallandale, Florida
  - Palm Beach Neurology - Premiere Research Institute, West Palm Beach, Florida
  - Neurostudies.net, Decatur, Georgia
  - Dekalb Neurology Associates, LLC, Lawrenceville, Georgia
  - NeuroStudies.net, Lawrenceville, Georgia
  - Clinical Research Institute, Wichita, Kansas
  - Monroe Community Hospital, Rochester, New York
  - Rhode Island Mood and Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Texas Neurology, P.A., Dallas, Texas
  - The Memory Clinic, Bennington, Vermont
  - University of Wisconsin, Department of Surgery, Madison, Wisconsin
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3133L1-2204&StudyName=Study%20Evaluating%20The%20Long-Term%20Safety%20And%20Efficacy%20Of%20Subcutaneous%20Bapineuzumab

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed the parent Study NCT00663026 and met the study criteria were enrolled and randomized into each of 3 dose cohorts to receive bapineuzumab or placebo. The study was terminated early on 06 August 2012 because 2 Phase 3 studies showed no clinical benefit. The decision was not based on any new safety concerns.
Groups:
- Bapineuzumab (5 mg + 5 mg): Participants who received 5 milligram (mg) in the parent study, in Study NCT00663026, continued to receive 5 mg bapineuzumab in the current study.
- Bapineuzumab (10 mg + 10 mg): Participants who received 10 mg in the parent study, Study NCT00663026, received 10 mg bapineuzumab in the current study.
- Placebo + Bapineuzumab 5mg: Participants who received placebo in the parent study, Study NCT00663026, received 5 mg bapineuzumab in the current study.
- Placebo + Bapineuzumab 10 mg: Participants who received placebo in the parent study, Study NCT00663026, received 10 mg bapineuzumab in the current study.
Period: Overall Study
Arm/Group | Bapineuzumab (5 mg + 5 mg) | Bapineuzumab (10 mg + 10 mg) | Placebo + Bapineuzumab 5mg | Placebo + Bapineuzumab 10 mg
Started | 24 | 21 | 10 | 7
Completed | 1 | 0 | 0 | 0
Not Completed | 23 | 21 | 10 | 7
Not completed — Adverse Event | 3 | 2 | 6 | 3
Not completed — Withdrawal by Subject | 3 | 2 | 0 | 1
Not completed — Caregiver Request | 3 | 2 | 1 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Discontinuation of Study by Sponsor | 8 | 13 | 3 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Other | 2 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study medication in study NCT00916617 were included in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bapineuzumab (5 mg + 5 mg) | Bapineuzumab (10 mg + 10 mg) | Placebo + Bapineuzumab 5mg | Placebo + Bapineuzumab 10 mg | Total
Number analyzed (Participants) | 23 | 21 | 10 | 7 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.2 (8.92) | 74.0 (9.34) | 80.4 (5.54) | 70.3 (10.13) | 73.9 (9.10)
Age, Customized [Number; unit: Participants]
  Less than (<) 65 years | 4 | 3 | 0 | 2 | 9
  Greater than or equal to (>=) 65 years | 19 | 18 | 10 | 5 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 6 | 2 | 30
  Male | 9 | 13 | 4 | 5 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Clinically Significant Magnetic Resonance Imaging (MRI) Findings
Description: A brain Magnetic Resonance Imaging (MRI) was obtained from all participants at Week 13 and quarterly thereafter. Participants were to meet the following criteria: screening brain MRI scan is consistent with the diagnosis of Alzheimer's Disease. Screening diagnosis of probable Alzheimer's disease according to National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria. Clinically significant MRIs were identified by the investigator. The number of participants with clinically significant MRIs are tabulated by visit and treatment group.
Time Frame: Week 13, 26, 39, 52, 65, 78, 91, 104, 117, 130, 143, 156, Any visit
Population: The safety population included all participants who received at least 1 dose of study medication in Study NCT00916617.
Measure: Number; unit: Participants
Arm/Group | Bapineuzumab (5 mg + 5 mg) | Bapineuzumab (10 mg + 10 mg) | Placebo + Bapineuzumab 5mg | Placebo + Bapineuzumab 10 mg
Number analyzed (Participants) | 23 | 21 | 10 | 7
Participants
  Week 13 | 0 | 2 | 1 | 0
  Week 26 | 1 | 0 | 1 | 0
  Week 39 | 0 | 0 | 0 | 0
  Week 52 | 0 | 0 | 0 | 0
  Week 65 | 0 | 0 | 0 | 0
  Week 78 | 0 | 1 | 0 | 0
  Week 91 | 0 | 0 | 0 | 0
  Week 104 | 0 | 0 | 0 | 0
  Week 117 | 0 | 0 | 0 | 0
  Week 130 | 0 | 0 | 0 | 0
  Week 143 | 0 | 0 | 0 | 0
  Week 156 | 0 | 0 | 0 | 0
  Any visit | 1 | 3 | 1 | 0

2. Secondary Outcome: Pharmacokinetic Parameters Including Maximal Serum Drug Concentration, Time to Maximal Serum Drug Concentration, and Terminal Half-life of Elimination
Time Frame: 36 months
Population: Because this study was terminated early, the planned pharmacokinetic analyses were not performed.
Arm/Group | Bapineuzumab (5 mg + 5 mg) | Bapineuzumab (10 mg + 10 mg) | Placebo + Bapineuzumab 5mg | Placebo + Bapineuzumab 10 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Bapineuzumab (5 mg + 5 mg) | Bapineuzumab (10 mg + 10 mg) | Placebo + Bapineuzumab 5mg | Placebo + Bapineuzumab 10 mg
Serious Adverse Events (participants affected / at risk) | 4/23 | 5/21 | 7/10 | 2/7
Other Adverse Events (participants affected / at risk) | 19/23 | 16/21 | 10/10 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bapineuzumab (5 mg + 5 mg) (N=23) | Bapineuzumab (10 mg + 10 mg) (N=21) | Placebo + Bapineuzumab 5mg (N=10) | Placebo + Bapineuzumab 10 mg (N=7)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bapineuzumab (5 mg + 5 mg) (N=23) | Bapineuzumab (10 mg + 10 mg) (N=21) | Placebo + Bapineuzumab 5mg (N=10) | Placebo + Bapineuzumab 10 mg (N=7)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 2 (2) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 2 (2) | 3 (4) | 1 (2) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (12) | 1 (3)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (9) | 4 (6) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 2 (5) | 1 (4)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (5) | 1 (1) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (8) | 2 (3) | 2 (3)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (6) | 2 (3) | 2 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Action tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Apraxia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Bradykinesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cogwheel rigidity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 2 (3) | 1 (1) | 1 (1) | 1 (1)
Dementia with Lewy bodies (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyporeflexia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Masked facies (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Movement disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sleep phase rhythm disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Vasogenic cerebral oedema (Nervous system disorders) | 3 (4) | 0 (0) | 2 (3) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cough (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysphonia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (2) | 2 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.